CLINICAL TRIAL: NCT01731769
Title: Preventing Seroma Formation After Axillary Lymph Node Dissection for Breast Cancer by Early Vacuum Assisted Closure--- a Randomized Control Clinical Trial
Brief Title: Preventing Seroma Formation After Axillary Lymph Node Dissection for Breast Cancer by Early Vacuum Assisted Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Bi-Hongda, attending physician,department of plastic surgery, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PSF-2012
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Breast Neoplasms
Keywords: Seroma Formation; Axillary Lymph Node Dissection; Breast cancer; Early Vacuum Assisted Closure
MeSH Terms: conditions — Breast Neoplasms | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Axillary dissection (Active Comparator): Axillary dissection is a surgical procedure that incises (opens) the armpit (axilla or axillary) to identify, examine, or remove lymph nodes (small glands, part of the lymphatic system, which filters cellular fluids).
  Interventions: Procedure: Axillary dissection
- vacuum assisted closure (Experimental): Vacuum assisted closure (also called vacuum therapy, vacuum sealing or topical negative pressure therapy) is a sophisticated development of a standard surgical procedure, the use of vacuum assisted drainage to remove blood or serous fluid from a wound or operation site.
  Interventions: Procedure: vacuum assisted closure in experimental arm

INTERVENTIONS:
Procedure: vacuum assisted closure in experimental arm
  Arms: vacuum assisted closure
Procedure: Axillary dissection
  Arms: Axillary dissection

SUMMARY:
Axillary dissection is the standard treatment for breast cancer patients with positive nodes. However, seroma formation after axillary dissection remains the most common early complication to breast cancer surgery. It can delay the initiation of adjuvant therapy, predispose to wound infection, delay wound healing and has also been linked to arm lymphoedema. Based on some studies and our experience that vacuum assisted closure （VAC）is effective in complex wound failures following axillary dissection and groin dissection, we use VAC to prevent seroma formation after extensive axillary dissection. This study is aimed to evaluate the efficacy, safety and economics benefits of early VAC application on postoperative complications and wound healing after extensive axillary dissection in comparison to conventional suction drain.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* patients diagnosed with breast cancer, receiving modified radical mastectomy and axillary dissection；
* Body Mass Index ≥28；
* drainage volume within the first 48 hours is more than 200 mL.

Exclusion Criteria:

* Subjects with coagulation disorders shown by exceeding the normal range of any of following: prothrombin time (PT), Quick, activated partial thromboplastin time (aPTT), fibrinogen level, or thrombocytes.
* Subjects having previously had axillary surgery,
* Subjects having undergone irradiation therapy to the axillary tissue
* Subjects having ever received chemotherapy before the surgery,
* Subjects with known hypersensitivity to components of the surgical sticky membrane

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
seroma formation complication incidence | within the first 30 days (plus or minus 3 days) after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China